CLINICAL TRIAL: NCT01254383
Title: An Open Label Crossover Study In Healthy Older Male Subjects To Evaluate The Pharmacokinetics And Safety Of Sildenafil Following Fasted Administration Of An Orally Disintegrating Tablet Formulation Of Sildenafil Administered With Or Without Water Relative To Viagra® Oral Tablet With Water
Brief Title: Pharmacokinetics Of Sildenafil Orally Disintegrating Tablet Formulation Versus To Viagra® Oral Tablet.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481289
Record Dates: First submitted 2010-11-19; First posted 2010-12-06 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: Bioequivalence Oral Dissolving Tablet
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator): Viagra 50 mg tablet, administered with approximately 240 mL water under fasted conditions
  Interventions: Drug: Sildenafil Tablet
- Treatment B (Experimental): Sildenafil ODT tablet 50 mg, administered without water under fasted conditions
  Interventions: Drug: Sildenafil ODT
- Treatment C (Experimental): Sildenafil ODT tablet 50 mg, administered with water under fasted conditions.
  Interventions: Drug: Sildenafil ODT

INTERVENTIONS:
Drug: Sildenafil Tablet — Tablet, 50 mg, Single Dose
  Arms: Treatment A
Drug: Sildenafil ODT — Orally Disintegrating Tablet, 50 mg, Single Dose
  Arms: Treatment B
Drug: Sildenafil ODT — Orally Disintegrating Tablet, 50 mg, Single Dose
  Arms: Treatment C

SUMMARY:
This study will evaluate if an orally disintegrating tablet of sildenafil will have similar pharmacokinetic properties as the conventional tablet of sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male subjects age 45 years or older with or without erectile dysfunction.

Body Mass Index (BMI) of 17.5 to 32.5 kg/m2.

Signed and dated informed consent document.

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities
* Have baseline orthostatic hypotension
* Positive drug screen, excessive alcohol and tobacco use

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) of sildenafil. | Up to 1 month
Cmax of sildenafil. | Up to 1 month

SECONDARY OUTCOMES:
AUC(0-inf) of sildenafil, if data permits. | Up to 1 month
Half-life of sildenafil, if data permits. | Up to 1 month
Tmax of sildenafil. | Up to 1 month
Number of patients with adverse events. | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- [Derived] Damle B, Duczynski G, Jeffers BW, Crownover P, Coupe A, LaBadie RR. Pharmacokinetics of a novel orodispersible tablet of sildenafil in healthy subjects. Clin Ther. 2014 Feb 1;36(2):236-44. doi: 10.1016/j.clinthera.2013.12.010. Epub 2014 Jan 18. PMID 24447534
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481289&StudyName=Pharmacokinetics%20Of%20Sildenafil%20Orally%20Disintegrating%20Tablet%20Formulation%20Versus%20To%20Viagra%AE%20Oral%20Tablet.%20%20